CLINICAL TRIAL: NCT06388811
Title: Validity and Reliability Study of the Turkish Version of the Early Osteoarthritis
Brief Title: Validity and Reliability Study of the Turkish Version of the Early Osteoarthritis Questionnaire
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fatma Merih Akpınar, Assistant Professor, Istanbul University
Other Study IDs: 2023/1162
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Early Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Knee Osteoarthritis Patients
  Interventions: Other: Early Osteoarthritis Questionnaire
- Population Without Knee Pain
  Interventions: Other: Early Osteoarthritis Questionnaire

INTERVENTIONS:
Other: Early Osteoarthritis Questionnaire — Self administered questionnaire

SUMMARY:
The symptoms of early osteoarthritis (OA) are quite similar to established knee OA, they differ, particularly in frequency, intensity, and severity. For this reason, in 2023, the International Symposium of intra-articular treatment (ISIAT) technical experts panel (TEP-technical experts panel) published for the first time a questionnaire designed to assess and monitor the follow-up and clinical progression of patients affected by early knee OA. Early management of knee OA is recommended by various guidelines because this approach may alter the course and clinical features of the disease, especially when considering disease-modifying agents that may delay disease progression.

Therefore, the assessment of early knee OA with a questionnaire may facilitate the follow-up of OA in the early stages of the disease when treatment is likely to be more effective. This approach will allow to reduce disability and improve patients' quality of life. While creating the Early Osteoarthritis Questionnaire (EOAQ), it was aimed to have a complete, short and easy-to-understand questionnaire and to ensure that the respondents could complete the questionnaire easily and in a short time. The EOAQ consists of 11 questions. The questions were divided into two different groups. While the first two questions were related with clinical characteristics, the other nine questions aimed to investigate the results reported by the patient. For each question, there are three responses depending on the number of episodes: Never, rarely (between one and three episodes) and frequently (more than three episodes) within a 6-month period. Turkish validity and reliability study of the EOAQ has not been conducted yet.

For the translation of the questionnaire, the guide recommended by Beaton et al. for the cultural adaptation of questionnaires will be used. According to this guideline the original EOAQ will be translated into Turkish by two experts independently of each other, and then a single Turkish version will be created by two experts working together. This Turkish version will then be translated back into English by an expert who can speak both languages at an advanced level. The experts will then evaluate the translation and adapt the questionnaire accordingly. After the completion of the translated form, 110 patients and 110 control group participants who applied to Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation and met the inclusion criteria will be included. The participants will be informed verbally and in writing about the purpose, duration and method of the study and will be asked to sign an "Informed Voluntary Consent Form" after their consent is obtained. Participants will fill in the Turkish version of the questionnaire. Along with the questionnaire, knee pain will be questioned with the Numeric Rating Scale (0=no pain, 10=the most severe pain you experience) and disability will be questioned with the WOMAC Questionnaire, whose Turkish validity and reliability study has been conducted. Test-retest method will be applied for reliability analyses; therefore, at least 30 patients among the patients included in the study will complete the questionnaire twice (the second evaluation will be 2 weeks after the first evaluation).

ELIGIBILITY:
Inclusion Criteria:

-

For the patient group :

1. Meeting the diagnostic criteria for early symptomatic knee OA

   * In the absence of risk factors, two mandatory symptoms (pain when climbing up and down stairs and increased pain with overload) are present
   * In the presence of 1 or 2 risk factors, at least pain when climbing up and down stairs is present among the two mandatory symptoms
   * Presence of at least 1 mandatory symptom in the presence of 3 or more risk factors
2. Over 40 years of age
3. Signing the informed consent form
4. Being able to read and write Turkish
5. To be able to come to the follow-ups required by the study

For the control group:

1. Absence of knee pain
2. Over 40 years of age
3. Signing the informed consent form
4. Being able to read and write Turkish
5. To be able to come to the follow-ups required by the study

Exclusion Criteria:

* For the patient group:

  1. Active inflammatory arthritis
  2. The presence of widespread pain
  3. Being under 40 years of age
  4. Having stage 1-4 knee OA according to Kellgren and Lawrence
  5. Recent trauma or injury
  6. Symptom duration of more than 6 months
  7. Having a mental capacity, cognition level that prevents understanding and completing the questionnaire

For the control group:

1. Having knee pain
2. Being under 40 years of age
3. Having a mental capacity, cognition level that prevents understanding and completing the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with early knee osteoarthritis and population without knee pain for control gorup
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2025-03-19 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Baseline, second week
  Patients rate their level of pain between 0-10 during movement, rest and night, 0 indicates no pain, 10 indicates the worst imaginable pain
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, second week
  WOMAC consists of 24 items consisting of 3 subgroups that the patients answer themselves. These subgroups include; pain intensity during various positions or movements, severity of joint stiffness and difficulty in performing daily functional activities. It has 3 forms: 5-point Likert, 100 mm visual analogue scale and 11-box numerical evaluation scale. The 5 point likert form will be filled in this study. Higher scores indicate worse pain, stiffness, or physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No